CLINICAL TRIAL: NCT03539627
Title: One-center, Observational, Non-interventional, Prospective Study of the Efficacy of Azilsartan Medoxomil in Patients With Arterial Hypertension Associated With Stable Ischemic Heart Disease and Type 2 Diabetes Mellitus.
Brief Title: Azilsartan Medoxomil in Hypertensive pAtients With Stable Ischemic Heart Disease and DiabEtes MEllitus.
Acronym: AcADEME
Status: Completed | Type: Observational
Sponsor: Research Institute for Complex Problems of Cardiovascular Diseases, Russia (Other)
Responsible Party: Principal Investigator, Olga Barbarash, Professor, Research Institute for Complex Problems of Cardiovascular Diseases, Russia
Other Study IDs: IISR-2017-102380
Record Dates: First submitted 2018-05-02; First posted 2018-05-29 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Arterial Hypertension; Diabetes Mellitus; Stable Chronic Angina
Keywords: diabetes mellitus; Edarbi; hypertension
MeSH Terms: conditions — Hypertension; Diabetes Mellitus; Angina, Stable | interventions — azilsartan medoxomil; Tablets; azilsartan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patients with hypertension, CAD and diabetes: Patients with hypertension associated with stable CAD and diabetes on azilsartan medoxomil (Edarbi) therapy
  Interventions: Drug: Azilsartan Medoxomil 40 MG Oral Tablet [Edarbi]

INTERVENTIONS:
Drug: Azilsartan Medoxomil 40 MG Oral Tablet [Edarbi] — patients are to receive azilsartan medoxomil

SUMMARY:
One-center, observational, non-interventional, prospective study of the efficacy of azilsartan medoxomil in patients with arterial hypertension associated with stable ischemic heart disease and type 2 diabetes mellitus.

DETAILED DESCRIPTION:
One-center, observational, non-interventional, prospective study of the efficacy of azilsartan medoxomil in patients with arterial hypertension associated with stable ischemic heart disease and type 2 diabetes mellitus.

During the study 5 visits to the research center are planned. At each visit, a physical examination, sampling of bio-samples for evaluation in the local laboratory, and collection of information on adverse events will be performed. 24-hours monitoring of blood pressure will be performed at screening, after 1 months of therapy and at the final visit (6 months of therapy).

Data will be collected during 5 consecutive visits to the research center. The observation period will be about 6 months, the active treatment period will be at least 6 months (24 weeks). Patients included in the study will be observed in an outpatient clinic according to the local practice of the research center.

It is planned that potentially eligible patients will be invited to the screening visit. Based on the results of daily monitoring of blood pressure, a final decision will be made about the suitability of the patient to participate in the study. Patients who have not reached the target values of blood pressure will start taking the study drug (Edarbi). By not achieving the target values of blood pressure, the mean daily systolic blood pressure is more than 130 mm Hg and the diastolic blood pressure is more than 90 mm Hg. The length of time between Visit 1 and Visit 2 is suspected to be no longer than 2 weeks.

All examinations (examination and evaluation of vital functions, laboratory tests, instrumental examinations) will be performed in accordance with the general standards of medical practice and in accordance with the routine practice of the institution.

Based on the number of patients hospitalized in the Research Institute For Complex Issues Of Cardiovascular Diseases (1500 patients), as well as the data on the prevalence of type 2 diabetes in this group (23.5%, 353 patients), the required sample size will be 184 patients (Confidence interval ± 5 %, the confidence probability is 95%).

SS = Z2 * (p) * (1-p) C2 where: Z = Z factor (1,96 for 95% confidence interval) p = percentage of respondents required, in decimal form (0,5 by default) c = confidence interval, in decimal form (for example, 0,04 = ±4%).

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent signed by the patient.
2. Men and women aged 18 years and older with a previously diagnosed hypertension and type 2 diabetes mellitus and stable ischemic heart disease.
3. Stable therapy of hypertension, T2DM and ischemic heart disease for at least 12 weeks before screening.
4. Not achievement of target values * of blood pressure against the background of previously prescribed and steadily accepted antihypertensive therapy.

   * not reaching the target figures of arterial pressure means mean systolic blood pressure more than 130 mm Hg and / or an average diastolic blood pressure more than 90 mmHg.
5. Investigator's decision on the advisability of correction of previously prescribed therapy with the replacement of ACE inhibitors or other ARBs with azilsartan medoxomil.

Exclusion Criteria:

1. Contraindications to the azilsartan medoxomil in accordance with instruction for use, including information on the individual intolerance of the drug.
2. Any circumstances in the opinion of the investigator that interfere with the participation of the patient in the study.
3. The patient included in the study is an employee of the center or a relative of the investigator.
4. Participation in other clinical trials. Participation in register studies is allowed.
5. Any disease or condition that leads to a decrease in the patient's life expectancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — adult patients only
Study Population: Patients with arterial hypertension associated with stable ischemic heart disease and type 2 diabetes mellitus
Sampling Method: Non-Probability Sample
Enrollment: 184 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2022-04-29 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure | interval: up to 24 weeks
  Dynamics of clinical SBP from the baseline against the background of therapy with Edarbi®

SECONDARY OUTCOMES:
Diastolic blood pressure | interval: up to 24 weeks
  Dynamics of clinical DBP from the baseline against the background of therapy with Edarbi® (interval: Visit of inclusion - Visit 5);
Dynamics of renal function (filtration) | interval: up to 24 weeks
  Dynamics of eGFR
Edarbi® efficacy | interval: up to 24 weeks
  proportion of patients who respond to Edarbi® therapy (defined as decrease of SBP≥ 20 mm Hg or decrease of DBP≥10 mm Hg)
Dynamics of renal function (evidence of kidney injury) | interval: up to 24 weeks
  N-GAL-dynamics
Dynamics of renal function (proteinuria detecton) | interval: up to 24 weeks
  UACR dynamics

CONTACTS AND LOCATIONS:
Locations (1):
- Anastasia Kochergina, Kemerovo, Russia

REFERENCES:
- See also: Kochergina A.M., Barbarash O.L. Azilsartan medoxomil: opportunities and prospects in diabetes mellitus. "Arterial'naya Gipertenziya" ("Arterial Hypertension"). 2021;27(2):247-254. (In Russ.) — https://htn.almazovcentre.ru/jour/article/view/2079